CLINICAL TRIAL: NCT02780986
Title: Efficacy of a Health Promotion and STI Prevention Program for Entertainment Establishments in Singapore
Brief Title: STI Prevention Program for Entertainment Establishments in Singapore
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government); National Skin Centre, Singapore (Other)
Responsible Party: Principal Investigator, Wong Mee Lian, Associate Professor, National University of Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDPHRG12NOV020
Record Dates: First submitted 2016-05-19; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Sexually Transmitted Infections
Keywords: female entertainment worker; heterosexual men; entertainment establishment; condom use; sexually transmitted infection; Singapore
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Female entertainment worker intervention group (Active Comparator): The intervention program for the female EE workers aims to increase STI/HIV prevention knowledge and develop their condom negotiation and application skills so as to increase condom use with both casual and paid partners. It consists of a total of 4 sessions: 2 on-site and 2 online sessions. For each on-site session, groups of 4 to 5 female EE workers will be gathered. The 2 on-site sessions would be delivered by peer educators. The 2 online sessions would be conducted via phone and other modes of network communication (e.g. SMS message or WhatsApp message) depending on the preference of each participant. In addition, all the intervention materials and video demonstrations will also be uploaded onto the web portal for the participant to access during their free time.
  Interventions: Behavioral: Female entertainment worker intervention group
- Female entertainment worker control group (No Intervention): The female EE workers in the control group will receive the same number of 2 onsite and 2 online sessions but covering healthy eating and physical activity.
  The following gives a summarised breakdown and content of each session:
  Session 1 (on-site immediately after baseline survey, 10 minutes):
  The peer educator will share information on healthy eating and physical activity using the educational pamphlets from the Health Promotion Board (HPB) with the participants.
  Session 2 (online 1-2 weeks after baseline survey, 5 minutes):
  The peer educator will share an app on healthy eating with the participants.
  Session 3 (online 3-4 weeks after baseline survey, 5 minutes):
  The peer educator will share an app on physical activity with the participants.
  Session 4 (onsite during follow-up survey, 10 minutes):
  The peer educator will reinforce information on healthy eating and physical activity based on the educational pamphlets from HPB with the participants.
- Heterosexual men intervention group (Active Comparator): The intervention program for heterosexual men patronising EEs will be a holistic non disease-centric, non-stigmatising and non-judgemental program addressing sexual well-being, avoidance of casual and paid sex if possible and safe sex such as condom use.
  Interventions: Behavioral: Heterosexual men intervention group
- Heterosexual men control group (No Intervention): There will be a simultaneous programme on healthy eating and physical activity at the control site at Tanjong Pagar. Health promoters will go around Tanjong Pagar and distribute pamphlets and brochures developed by the HPB on healthy eating and physical activity to the heterosexual men who step into or out of the EEs there. These health promoters have been trained to give simple health advice on healthy eating and physical activity if the heterosexual men wish to find out more information.

INTERVENTIONS:
Behavioral: Female entertainment worker intervention group — The following summarises the content of each session:
  Session 1 (on-site): The peer educator will play 2 videos, demonstrating 5 sexy ways of putting on a condom in a pleasurable manner, and another one focusing on condom negotiation skills.
  Session 2 (online): The peer educator will share an app game on condom usage and relevant online resources with the participants.
  Session 3 (onsite): There will be discussion of common problems encountered in condom usage and condom negotiation by the participants. The peer educators will then conduct role plays with the participants to demonstrate the counter-strategies. In addition, the peer educators will get the participants who have been successful in condom negotiation to share their success stories.
  Session 4 (online): The peer educator will share information about safe consumption of alcohol and tips to avoid getting drunk through the online platforms.
  Arms: Female entertainment worker intervention group
Behavioral: Heterosexual men intervention group — This will be delivered via 3 main activities:
  1. Edutainment in the form of talk-shows based on 6 themes of sexual well-being and safe sex, held in the EE setting hosted by a famous female local comedian.
  2. Web portal named THINK: This contains educational materials based on 6 themes of sexual health and safe sex, HIV risk profiling tool to calculate the risk of contracting HIV, videos on true life experiences of heterosexual men engaging in high risk sexual behaviour and another video on exit strategies to avoid casual or paid sex, online support for STI testing services and consultation with a clinical sexologist.
  3. Public education event/photo booth: i. Distribution of pamphlets and brochures on sexual well-being and safe sex ii. Interactions with health promoters iii. Photo taking on safe sex messages iv. Free access to condoms and lubricants
  Arms: Heterosexual men intervention group

SUMMARY:
The investigators aim to assess the efficacy of a multi-component intervention on condom use and sexually transmitted infection (STIs) in female entertainment workers and men frequenting entertainment establishments (EEs), using a quasi-experimental design. Joo Chiat and Golden Mile Complex will be selected purposively as control cluster sites (n=220) with follow-up of entertainment workers at 6 weeks. The same sites will be used as intervention sites after a 3-months 'wash out' period. Self-reported condom use, vaginal swab samples for polymerase chain reaction (PCR) for cervical gonorrhoea and chlamydia infections, and throat swabs for culture for pharyngeal gonorrhoea will be assessed. Clark Quay will be the intervention venue for the heterosexual men while Tanjong Pagar will be the equivalent control site. Using time location sampling, cross-sectional samples of men patronising these establishments will be assessed on self-reported condom use at baseline (n=600) and 6 months after the intervention (n=400) in both intervention and control groups.

DETAILED DESCRIPTION:
BACKGROUND:

Globalisation has led to an influx of women from surrounding Asian countries with high prevalence of sexually transmitted infections (STIs) to work in entertainment establishments (EEs) in Singapore. Men frequenting EEs reported high levels of unprotected sex with commercial and casual partners.

OBJECTIVES:

The aim is to assess the efficacy of a multi-component intervention on STI prevention and condom use in female entertainment workers and men frequenting EEs in Singapore, using a quasi-experimental design. The hypothesis is that a comprehensive sexual health promotion program which incorporates behavioural (STI/HIV education, condom use and condom negotiation skills), biomedical (STI screening and treatment services) and structural components (free access to condoms) to female entertainment workers as well as behavioural (sexual well-being and safe sex edutainment) and structural (free access to condoms) interventions to men patronising EEs in Singapore will achieve an increase in condom use (for both target groups) and a reduction in incident STIs (only for female EE workers).

METHODS:

Female EE workers:

Joo Chiat and Golden Mile Complex will be selected purposively as control cluster sites with 220 entertainment workers being recruited and followed up at 6 weeks. The same sites will be used as intervention sites with recruitment of a separate sample of 220 participants after a 3-months' 'wash out' period to ensure comparability. Self-reported condom use, vaginal swab samples for polymerase chain reaction (PCR) for cervical gonorrhoea and chlamydia infections, and throat swabs for culture for pharyngeal gonorrhoea will be assessed. The short follow-up period is because almost all of these women come to Singapore to work illegally on 1 to 2 months social visit passes.

Heterosexual men:

The investigators are unable to recruit heterosexual men from the same study sites of the female EE workers due to feasibility and safety considerations. Instead, Clark Quay will be selected purposively as the intervention site for the heterosexual men. Tanjong Pagar will be the equivalent control site. Using time location sampling, cross-sectional samples of men patronising these establishments will be assessed on self-reported condom use at baseline (n=600) and 6 months after the intervention (n=400) in both intervention and control groups.

MAIN OUTCOMES:

The primary outcomes for female EE workers are consistent condom use for vaginal sex with paid and casual partner respectively in the past 1 month and the secondary outcome is STI incidence. The primary outcomes for heterosexual men are condom use at last vaginal and oral sex respectively with casual partner in the past 6 months.

POSSIBLE APPLICATIONS:

The study will provide pertinent data for planning STI/HIV prevention programs for female entertainment workers and men patronising EEs in Singapore and the region.

ELIGIBILITY:
Inclusion Criteria:

For female EE workers:

Female entertainment worker who is either a Vietnamese or Thai between the ages of 18 to 69 years old satisfying the 2 criteria:

(i) Planning to work for at least 6 weeks after the baseline survey in Singapore (ii) Have engaged in vagina, oral or anal sex with either a casual or paid male partner in the past month

The casual or paid male partner need not come from the EE that the female EE worker works in.

For heterosexual men:

Male resident who is either a Singapore Citizen or a Permanent Resident between the ages of 21 to 69 years satisfying the 2 criteria:

(i) Patronise the EEs in the site at least once in the past 6 months (ii) Have engaged in vagina, oral or anal sex with either a casual or paid female partner in the past 6 months

The casual or paid female partner need not come from the EEs in the site that the heterosexual man has patronised.

Exclusion Criteria:

For female EE workers in the intervention group only:

Female EE workers who have participated in the control group would be excluded from participating in the intervention group

For heterosexual men during the post-intervention survey of the control group only:

Heterosexual men from the control site who have patronised EEs in the intervention site or who have been exposed to the interventions in the past 6 months would be excluded from the post-intervention survey for the control group.

For heterosexual men during the post-intervention survey of the intervention group only:

Heterosexual men from the intervention site who have not been exposed to at least 1 of the 3 main activities of the intervention in the past 6 months would be excluded from the post-intervention survey for the intervention group.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Consistent condom use for vaginal sex with paid partners (for female entertainment workers) | 1 month
  This is assessed by 2 questions, "Did the participant ever have vaginal sex in the past 1 month?" (Options of no and yes) and "If the participant had vaginal sex, how often did she use condoms with paid partners?" (Options of not applicable, never, sometimes and always). Participants who give the answer as 'Yes' to the first question and 'Always' to the second question are classified as having consistent condom usage for vaginal sex with paid partners.
Consistent condom use for vaginal sex with casual partners (for female entertainment workers) | 1 month
  This is assessed by 2 questions, "Did the participant ever have vaginal sex in the past 1 month?" (Options of no and yes) and "If the participant had vaginal sex, how often did she use condoms with casual partners?" (Options of not applicable, never, sometimes and always). Participants who give the answer as 'Yes' to the first question and 'Always' to the second question are classified as having consistent condom usage for vaginal sex with causal partners.
Condom use at last vaginal sex with casual partners (for heterosexual men) | 6 months
  This is determined by 2 questions, "Did the participant ever have vaginal sex in the past 6 months?" (Options of no and yes) and "If the participant had vaginal sex, did he use a condom the last time he had vaginal sex with the casual partner?" (Options of not applicable, no and yes). Participants who give the answer as 'Yes' to the first question and 'Yes' to the second question are classified as having used condom at last vaginal sex with casual partners.
Condom use at last oral sex with casual partners (for heterosexual men) | 6 months
  This is determined by 2 questions, "Did the participant ever have oral sex in the past 6 months?" (Options of no and yes) and "If the participant had oral sex, did he use a condom the last time he had oral sex with the casual partner?" (Options of not applicable, no and yes). Participants who give the answer as 'Yes' to the first question and 'Yes' to the second question are classified as having used condom at last oral sex with casual partners.

SECONDARY OUTCOMES:
STI incidence (for female entertainment workers) | 6 weeks
  This is defined as having a positive laboratory test result for a new episode of cervical chlamydia, cervical gonorrhoea or pharyngeal gonorrhoea at 6 weeks post-intervention.
Consistent condom use for oral sex with paid partners (for female entertainment workers) | 1 month
Consistent condom use for oral sex with casual partners (for female entertainment workers) | 1 month
Consistent condom use for vaginal sex with casual partners (for heterosexual men) | 6 months
HIV knowledge (for both target groups) | 1 month for female entertainment workers and 6 months for heterosexual men
Success in condom negotiation (for female entertainment workers) | 1 month
Number of sexual partners (for both target groups) | 1 month for female entertainment workers and 6 months for heterosexual men
HIV/STI testing uptake (for heterosexual men) | 6 months
Consistent and last condom use with regular partners (for both target groups) | 1 month for female entertainment workers and 6 months for heterosexual men
Consistent condom use for oral sex with casual partners (for heterosexual men) | 6 months
Consistent and last condom use with female entertainment workers (for heterosexual men) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mee Lian Wong, MBBS, MPH, MD, Principal Investigator — Saw Swee Hock School of Public Health, National University of Singapore
Locations (1):
- Saw Swee Hock School of Public Health, National University of Singapore, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Wong ML, Chan R, Tan HH, Yong E, Lee L, Cutter J, Tay J, Koh D. Sex work and risky sexual behaviors among foreign entertainment workers in urban Singapore: findings from Mystery Client Survey. J Urban Health. 2012 Dec;89(6):1031-44. doi: 10.1007/s11524-012-9723-5. PMID 22707309
- [Background] Wong ML, Chan KW, Koh D. A sustainable behavioral intervention to increase condom use and reduce gonorrhea among sex workers in Singapore: 2-year follow-up. Prev Med. 1998 Nov-Dec;27(6):891-900. doi: 10.1006/pmed.1998.0398. PMID 9922072
- [Background] Wong ML, Chan R, Koh D. Long-term effects of condom promotion programmes for vaginal and oral sex on sexually transmitted infections among sex workers in Singapore. AIDS. 2004 May 21;18(8):1195-9. doi: 10.1097/00002030-200405210-00013. PMID 15166535
- [Background] Chan R, Goh CL. STD/AIDS knowledge and risk behaviour among masseuses and bar hostesses in Singapore. Int J STD AIDS. 1997 Jun;8(6):373-7. doi: 10.1258/0956462971920280. PMID 9179647
- [Background] Heng BH, Lee HP, Kok LP, Ong YW, Ho ML. A survey of sexual behaviour of Singaporeans. Ann Acad Med Singap. 1992 Nov;21(6):723-9. PMID 1295409
- [Background] Sen P, Chio MT, Tan HH, Chan RK. Rising trends of STIs and HIV infection in Singapore-- a review of epidemiology over the last 10 years (1994 to 2003). Ann Acad Med Singap. 2006 Apr;35(4):229-35. PMID 16710492
- [Derived] Lim RBT, Tham DKT, Cheung ON, Adaikan PG, Wong ML. A Public Health Communication Intervention Using Edutainment and Communication Technology to Promote Safer Sex among Heterosexual Men Patronizing Entertainment Establishments. J Health Commun. 2019;24(1):47-64. doi: 10.1080/10810730.2019.1572839. Epub 2019 Jan 30. PMID 30698082
- [Derived] Lim RBT, Cheung ONY, Tham DKT, La HH, Win TT, Chan R, Wong ML. Using qualitative and community-based engagement approaches to gain access and to develop a culturally appropriate STI prevention intervention for foreign female entertainment workers in Singapore. Global Health. 2018 Apr 16;14(1):36. doi: 10.1186/s12992-018-0358-5. PMID 29661249
- [Derived] Lim RB, Wong ML, Cheung ON, Tham DK, Tai BC, Chan R. Factors associated with consistent condom use and STIs among foreign female entertainment workers: results from a cross-sectional survey in Singapore. Sex Transm Infect. 2017 Mar;93(2):118-124. doi: 10.1136/sextrans-2015-052530. Epub 2016 Jul 7. PMID 27388458